CLINICAL TRIAL: NCT03388411
Title: Nutritional Intake, Metabolic Abnormalities and Gut Microbiome in Children
Brief Title: Nutritional Intake and Gut Microbiome
Status: Completed | Type: Observational
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ky Young Cho, Clinical Professor, Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: Gut microbiome
Record Dates: First submitted 2017-12-19; First posted 2018-01-03 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Obesity, Childhood
Keywords: Microbiome; Gut
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese children: Children ≥95 ‰ between age 7 and 12 years
  Interventions: Diagnostic Test: Gut microbiome profiling
- Non-obese children: 5‰< BMI <85 ‰ for children between the ages of 7 and 12 years
  Interventions: Diagnostic Test: Gut microbiome profiling

INTERVENTIONS:
Diagnostic Test: Gut microbiome profiling — Gut microbial profiling will be done with next-generation sequencing targeting bacterial 16s rRNA genes.
  Other Names: 16s metagenomic analysis

SUMMARY:
Pediatric obesity has been increasing in prevalence, but concerns have been raised around the world because no treatment has been found. Recently, however, research on gut microbiome has begun to become a new alternative. It has been shown that changes in the microbiome in adults may induce obesity. However, the results on children are still scarce. Unlike adults, children have few external factors such as alcohol, tobacco, stress, and cancer, making them suitable for obesity-related gut microbiome studies. The investigators will use Illumina MiSeq platform for 16s rRNA metagenomics profiling in children. In this study, the investigators aimed to analyze the relationship between pediatric obesity, gut microbiome profile, blood biomarkers relevant to metabolic syndrome, and nutrient intake data.

ELIGIBILITY:
Inclusion Criteria:

* Obese children: Children ≥95 ‰ between age 7 and 12 years
* Non-obese children: 5‰<BMI <85 ‰ for children between the ages of 7 and 12 years

Exclusion Criteria:

* Taking antibiotics, probiotics, or steroids for a month before visit
* Taking probiotics-like products including yogurt for seven days before visit
* Having enteritis symptoms including diarrhea for a month before visit
* Chronic heart disease, chronic bowel disease, chronic liver disease, chronic kidney disease, endocrine disease, genetic diseases or congenital metabolic disorder

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary care clinic and community samples
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Correlation of fecal microbial profile with childhood obesity | visit 1day
  Analysis of fecal microbial profile using 16s rRNA sequencing
Correlation of fecal microbial profile with nutrient intake data using feeding diary | visit 1day
  Nutritional intake analysis of total calorie, carbohydrate, fiber, fat, and protein from feeding dairy for two days

SECONDARY OUTCOMES:
Correlation of childhood obesity with metabolic abnomalities using blood sampling | visit 1day
  Glucose, AST, ALT, uric acid, triglyceride, HDL-cholesterol, LDL-cholesterol, total cholesterol, insulin, hsCRP, 25(OH)-Vitamin D3, hemoglobin, ferritin, and HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Ky Young Cho, M.D., Principal Investigator — Kangnam Sacred Heart Hospital, Hallym University College of Medicine
Locations (1):
- Hallym University Kangnam Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Study participants will only agree if IPD is not shared.

REFERENCES:
- [Background] Clemente JC, Ursell LK, Parfrey LW, Knight R. The impact of the gut microbiota on human health: an integrative view. Cell. 2012 Mar 16;148(6):1258-70. doi: 10.1016/j.cell.2012.01.035. PMID 22424233
- [Background] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603
- [Background] Eckburg PB, Bik EM, Bernstein CN, Purdom E, Dethlefsen L, Sargent M, Gill SR, Nelson KE, Relman DA. Diversity of the human intestinal microbial flora. Science. 2005 Jun 10;308(5728):1635-8. doi: 10.1126/science.1110591. Epub 2005 Apr 14. PMID 15831718
- [Background] Yun Y, Kim HN, Kim SE, Heo SG, Chang Y, Ryu S, Shin H, Kim HL. Comparative analysis of gut microbiota associated with body mass index in a large Korean cohort. BMC Microbiol. 2017 Jul 4;17(1):151. doi: 10.1186/s12866-017-1052-0. PMID 28676106
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Hu HJ, Park SG, Jang HB, Choi MK, Park KH, Kang JH, Park SI, Lee HJ, Cho SH. Obesity Alters the Microbial Community Profile in Korean Adolescents. PLoS One. 2015 Jul 31;10(7):e0134333. doi: 10.1371/journal.pone.0134333. eCollection 2015. PMID 26230509
- [Background] Cox AJ, West NP, Cripps AW. Obesity, inflammation, and the gut microbiota. Lancet Diabetes Endocrinol. 2015 Mar;3(3):207-15. doi: 10.1016/S2213-8587(14)70134-2. Epub 2014 Jul 22. PMID 25066177
- [Background] Schwiertz A, Taras D, Schafer K, Beijer S, Bos NA, Donus C, Hardt PD. Microbiota and SCFA in lean and overweight healthy subjects. Obesity (Silver Spring). 2010 Jan;18(1):190-5. doi: 10.1038/oby.2009.167. Epub 2009 Jun 4. PMID 19498350
- [Background] Turnbaugh PJ, Backhed F, Fulton L, Gordon JI. Diet-induced obesity is linked to marked but reversible alterations in the mouse distal gut microbiome. Cell Host Microbe. 2008 Apr 17;3(4):213-23. doi: 10.1016/j.chom.2008.02.015. PMID 18407065
- [Background] Jumpertz R, Le DS, Turnbaugh PJ, Trinidad C, Bogardus C, Gordon JI, Krakoff J. Energy-balance studies reveal associations between gut microbes, caloric load, and nutrient absorption in humans. Am J Clin Nutr. 2011 Jul;94(1):58-65. doi: 10.3945/ajcn.110.010132. Epub 2011 May 4. PMID 21543530
- [Background] Pedersen HK, Gudmundsdottir V, Nielsen HB, Hyotylainen T, Nielsen T, Jensen BA, Forslund K, Hildebrand F, Prifti E, Falony G, Le Chatelier E, Levenez F, Dore J, Mattila I, Plichta DR, Poho P, Hellgren LI, Arumugam M, Sunagawa S, Vieira-Silva S, Jorgensen T, Holm JB, Trost K; MetaHIT Consortium; Kristiansen K, Brix S, Raes J, Wang J, Hansen T, Bork P, Brunak S, Oresic M, Ehrlich SD, Pedersen O. Human gut microbes impact host serum metabolome and insulin sensitivity. Nature. 2016 Jul 21;535(7612):376-81. doi: 10.1038/nature18646. Epub 2016 Jul 13. PMID 27409811
- [Background] Yoo JY, Kim SS. Probiotics and Prebiotics: Present Status and Future Perspectives on Metabolic Disorders. Nutrients. 2016 Mar 18;8(3):173. doi: 10.3390/nu8030173. PMID 26999199
- [Background] Fadrosh DW, Ma B, Gajer P, Sengamalay N, Ott S, Brotman RM, Ravel J. An improved dual-indexing approach for multiplexed 16S rRNA gene sequencing on the Illumina MiSeq platform. Microbiome. 2014 Feb 24;2(1):6. doi: 10.1186/2049-2618-2-6. PMID 24558975